CLINICAL TRIAL: NCT00176657
Title: Comparison of Whole Blood Return and Normal Practice Red Blood Cell Salvage Return Following Cardiopulmonary Bypass
Brief Title: The Use of HEMOBAG to Salvage Blood After Cardiac Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inability to attain sufficient numbers of subjects
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: Global Blood Resources, LLC (Other)
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0120040166
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2007-05-01 (Estimated); Status verified 2007-04

CONDITIONS: Cardiopulmonary Bypass; Cardiac Diseases
Keywords: cardiac surgery; transfusion
MeSH Terms: conditions — Heart Diseases

INTERVENTIONS:
Drug: HEMOBAG Assessment

SUMMARY:
The avoidance of blood transfusions benefits the patient. Cardiopulmonary bypass (CPB) is routinely used in complex cardiac surgeries. This device requires circulating blood through an oxygenator and pump while the heart is stopped. Upon discontinuation of CPB, the volume of blood in the CPB circuit, approximately 1 to 1.5 liters, is currently processed for the red cell components of the blood. Yet, all the other blood components are available in this volume of blood, but are discarded. The Hemobag filters allow for whole blood reinfusion rather than just red cell reinfusion. Thus, the patient's own platelets, for example, are returned to the patient. The product is just being used clinically and we, the investigators at University of Medicine and Dentistry, New Jersey, have been asked to perform a study on our normal practice (red blood cell return as described above) compared to the whole blood return available with the Hemobag™.

DETAILED DESCRIPTION:
The HemobagTM is a bag containing a microfilter for separation of autologous whole blood from intravenous solutions to provide a whole blood reinfusion from a cardiopulmonary bypass machine.

Following cardiopulmonary bypass (CPB), blood remaining within the bypass machine circuit is normally processed by a centrifugal separation of fluids from red blood cells (RBCs) and the RBCs are reinfused back into the patient. An FDA approved device, the HemobagTM, provides an alternative by reinfusing whole blood, including RBCs, from the CPB machine circuit. This allows the patient's own whole blood to be returned back to the patient with all components including functioning, non-activated platelets, coagulation factors and plasma. In preliminary human trials, blood measurements were improved in patients whose CPB blood was processed through the HemobagTM.

This study will evaluate 50 patients whose post-CPB blood is processed by normal practice (centrifugal separation of RBCs for reinfusion) or HemobagTM whole blood reinfusion. Outcome measurements will be chest tube drainage for the initial 24 hours following on-pump cardiac surgery, ventilatory requirements, protein levels, transfusion requirements, coagulation profile, A/A gradients, arterial blood gas measures, and CBC blood panels. All of these data are available from the normal clinical care of the patient.

The hypothesis is that the HemobagTM treated patients will have improved physiologic function from the return of whole blood rather than just RBCs following cardiac surgery using CPB.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between the ages of 18 and 80 years of age, who are mentally capable of giving an informed consent.
* Electively scheduled cardiac or open heart surgery using the cardiopulmonary bypass pump.

Exclusion Criteria:

* Failure to provide an informed consent
* History of trans ischemic attacks (TIA) and/or stroke with residual neurological or cognitive dysfunction
* Currently on dialysis (treatment for kidneys with little or no function)
* History of impaired liver function or coagulopathy
* Hemodynamic instability, cardiogenic shock or severe cardiomegaly
* Scheduled combined surgical procedure (i.e. coronary artery bypass graft [CABG] and endarterectomy)
* If patient has received more than two units of blood in the 12 hours preceding randomization.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-09; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Hematology value
Days of hospital stay

SECONDARY OUTCOMES:
Patient's morbidity
Complication rate

CONTACTS AND LOCATIONS:
Overall Officials: Douglas J Jackson, MD, Principal Investigator — UMDNJ Dept. of Anesthesiology
Locations (1):
- UMDNJ, Newark, New Jersey, United States